CLINICAL TRIAL: NCT05291195
Title: Treatment of Chronic Periapical Periodontitis of Young Permanent Teeth by Means of Three Adjuvant Treatment Approaches: A Prospective Comparative Microbiological and Clinical Study
Brief Title: Treatment of Young Permanent Teeth With Different Adjuvant Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Dragana Rakasevic, Principal Investigator and Research Associate, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36/7
Record Dates: First submitted 2022-02-17; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-01

CONDITIONS: Treatment; Periodontitis, Apical; Necrotic Pulp
Keywords: young permanent teeth; periodontitis apical; treatment
MeSH Terms: conditions — Periapical Periodontitis; Dental Pulp Necrosis | interventions — Lasers; Oils, Volatile

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Laser-devices group (Experimental): Mechanico-chemical root canal preparation and root canal disinfection were be performed by means of mechanic-chemical methods including hand instruments followed by 1.5% sodium hypochlorite. Afterwards, depending on allocations, in the laser devices group, adjuvant treatment approaches were be performed by means of laser devices either photodynamic therapy (HELBO, Photodynamic Systems GmbH), or high power diode laser (940nm, Biolase).
  Interventions: Device: Laser-device group; Drug: Sodium hypochlorite group
- Sodium hypochlorite (Experimental): Mechanico-chemical root canal preparation and root canal disinfection were be performed by means of mechanic-chemical methods including hand instruments followed by 1.5% sodium hypochlorite (pH 12), at room temperature (21 degrees Celsius).
  Interventions: Drug: Sodium hypochlorite group
- Essential oil (Experimental): Mechanico-chemical root canal preparation and root canal disinfection were be performed by means of mechanic-chemical methods including hand instruments followed by 1.5% sodium hypochlorite (pH 12), at room temperature (21 degrees Celsius).
  Depending on allocations, in the essential oil group, the canals were be treated with adjuvant essential oil of Cymbopogon martinii and Thymus vulgaris (Herba oils, Herba doo, Belgrade, Serbia)
  Interventions: Drug: Essential Oil; Drug: Sodium hypochlorite group

INTERVENTIONS:
Device: Laser-device group — After each instrumentation, the root canals were irrigated with 1.5 % sodium hypochlorite (NaOCl).
  Depending on allocations, in the laser-device groups, the adjuvant treatment approaches were performed either by means of photodynamic therapy (HELBO, Photodynamic Systems GmbH) or high power diode laser (940nm, Biolase ® Technology, CA, USA). Performing photodynamic therapy the root canals were filled with the phenothiazine chloride (HELBO® Endo Blue, Bredent, Germany) for 2 min following irradiation of diode laser (HELBO® TheraLite Laser (λ = 660 nm, power = 100 mW)) for 60 s. Performing only diode laser the root canals were be irrigated with a diode laser (λ = 940 maximal power 10W) for 60 s.
  Other Names: Laser
  Arms: Laser-devices group
Drug: Essential Oil — After each instrumentation, the root canals were irrigated with 1.5 % sodium hypochlorite (NaOCl).
  Depending on allocations, in the EO group, the adjuvant treatment approaches were performed either by means of essential oil (Cymbopogon martinii and Thymus vulgaris, Herba oils, Herba d.o.o, Belgrade, Serbia)
  Other Names: EO
  Arms: Essential oil
Drug: Sodium hypochlorite group — Mechanico-chemical root canal preparation and root canal disinfection were be performed by means of mechanic-chemical methods including hand instruments followed by 1.5% sodium hypochlorite (pH 12), at room temperature (21 degrees Celsius).
  Other Names: NaOCl group

SUMMARY:
To determine microbiology assessment of infected root canal in young permanent teeth, as well as antimicrobial efficiency of different adjuvant treatment modalities including photodynamic therapy (PDT), high-power diode laser, and essential oils following mechanic-chemical treatment in the treatment of periapical periodontitis in these teeth.

DETAILED DESCRIPTION:
To determine antimicrobial efficiency of adjuvant photodynamic therapy (PDT) and high-power diode laser, and essential oils in the treatment of chronic periapical periodontitis in young permanent teeth.

Material and Methods: Young permanent teeth with chronic periapical periodontitis were selected and randomly divided into tests and control groups. Adjuvant treatment approaches were randomly performed following standard mechanical-chemical endodontic treatment:

1. Experimental laser-device 1, PDT group: adjuvant PDT (n=10)
2. Experimental laser-device 2, Diode laser (940 nm, 1W) (n=10)
3. Experimental essential oil (n=10)
4. Experimental sodium hypochlorite (NaoCL) group (n= 10) solely mechanical instrumentation with 1.5 % of NaOCl irrigation was performed (positive control).

Afterwards, each root canal was filled with calcium hydroxide, and definitive obturation was done seven days respectively.

Microbiological analyses of root canals were assessed after accessing the canal (sample 1), following mechanical-chemical treatment (sample 2), and adjuvant treatment approaches (sample 3). The microbiological identification and quantification were provided by MALDI -TOF spectrometry and plate count assay. To evaluate the efficiency of treatment modalities, radiography records were additionally used.

ELIGIBILITY:
Inclusion Criteria:

* Had signed informed consent by the parents or legal guardian ;
* Systemically healthy children;
* Had not been submitted to antibiotic therapy in the previous 3 months;
* Had a least one young permanent anterior tooth (incisor or canine) or the first premolar with pulp necrosis and presence of a chronic periapical lesion (CPP);
* Had no endodontic treatment of the selected tooth;
* Had no signs of an acute condition;

Exclusion Criteria:

* Presence of systemic diseases such as diabetes mellitus, asthma, chronic infections, immunosuppressive diseases or other that could compromise the patient immune system
* Use anti-inflammatory or immunosuppressive therapy in the last 6 months;
* Patients with antibiotic prophylactic requirements before dental treatment;

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Number of teeth without bacteria load after laser-devices and essential oil in endodontic treatment | 6 months
  The number of teeth without isolated bacteria load were assessed. Microbiological samples from the root canals were collected immediately after accessing the canal, following endodontic treatment, and after the adjuvant treatments in allocated groups (Photodynamic therapy or Diode laser or Essential oil). The microbiological identification and quantification were provided by MALDI -TOF spectrometry and plate count assay.
Number of teeth without bacteria load after sodium hypochlorite (NaOCl) in endodontic treatment | 6 months
  The number of teeth without isolated bacteria load were assessed after sodium hypochlorite irrigation in each group (Laser-device, Essential oil and Sodium hypochlorite). Microbiological samples from the root canals were collected immediately after accessing the canal, following the endodontic treatment. The microbiological identification and quantification were provided by MALDI -TOF spectrometry and plate count assay.

SECONDARY OUTCOMES:
Radiography record of periapical lesion healing | Change baseline radiography record at 6 months
  Radiography record of periapical lesion taken by parallel long cone beam technique

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Markovic, Professor, Study Chair — University of Zagreb
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Gained results are planned to be published in international journals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 2022. to 2032.
Access Criteria: The investigators will be shared analyzed outcomes and procedure protocols, as well as microbiological analyses methods.

REFERENCES:
- [Background] Banchs F, Trope M. Revascularization of immature permanent teeth with apical periodontitis: new treatment protocol? J Endod. 2004 Apr;30(4):196-200. doi: 10.1097/00004770-200404000-00003. PMID 15085044
- [Background] Mohammadi Z, Jafarzadeh H, Shalavi S, Yaripour S, Sharifi F, Kinoshita JI. A Review on Triple Antibiotic Paste as a Suitable Material Used in Regenerative Endodontics. Iran Endod J. 2018 Winter;13(1):1-6. doi: 10.22037/iej.v13i1.17941. PMID 29692827
- [Background] Yun KH, Lee HS, Nam OH, Moon CY, Lee JH, Choi SC. Analysis of bacterial community profiles of endodontically infected primary teeth using pyrosequencing. Int J Paediatr Dent. 2017 Jan;27(1):56-65. doi: 10.1111/ipd.12226. Epub 2016 Feb 12. PMID 26872127
- [Background] Cheng X, Guan S, Lu H, Zhao C, Chen X, Li N, Bai Q, Tian Y, Yu Q. Evaluation of the bactericidal effect of Nd:YAG, Er:YAG, Er,Cr:YSGG laser radiation, and antimicrobial photodynamic therapy (aPDT) in experimentally infected root canals. Lasers Surg Med. 2012 Dec;44(10):824-31. doi: 10.1002/lsm.22092. Epub 2012 Nov 20. PMID 23168798
- [Background] Marinkovic J, Culafic DM, Nikolic B, Dukanovic S, Markovic T, Tasic G, Ciric A, Markovic D. Antimicrobial potential of irrigants based on essential oils of Cymbopogon martinii and Thymus zygis towards in vitro multispecies biofilm cultured in ex vivo root canals. Arch Oral Biol. 2020 Sep;117:104842. doi: 10.1016/j.archoralbio.2020.104842. Epub 2020 Jul 16. PMID 32707220